CLINICAL TRIAL: NCT00315055
Title: Immunogenicity of DTaP-IPV-Hep B-PRP~T Combined Vaccine Compared With PENTAXIM™ and ENGERIX B® at 2, 3, and 4 Months Primary Schedule in Healthy Turkish Infants
Brief Title: Immunogenicity of DTaP-IPV-Hep B-PRP~T Combined Vaccine Compared With PENTAXIM™ and ENGERIX B® at 2-3-4 Months Schedule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L10
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis B; Polio; Diphtheria; Pertussis
Keywords: Hepatitis B; Polio; Diphtheria; Pertussis; H influenzae type b
MeSH Terms: conditions — Hepatitis B; Poliomyelitis; Diphtheria; Whooping Cough; Haemophilus Infections | interventions — DTaP-IPV-HB-PRP-T vaccine; Pentavac; Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: DTaP-IPV-Hep B-PRP-T (Experimental): Participants will receive 3 vaccinations with Diphtheria (D) and tetanus (T) toxoids, acellular pertussis (2-component) (aP), recombinant Hepatitis B surface antigen (HBsAg), inactivated poliomyelitis virus (IPV), and Hemophilus influenzae type b (Hib) polysaccharide conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T); One dose each at 2, 3, and 4 months of age.
  Interventions: Biological: DTaP-IPV-HB-PRP~T vaccine
- Group 2: PENTAXIM™ and ENGERIX B® PEDIATRIC (Active Comparator): Participants will receive 3 vaccinations with DTaP-IPV-PRP~T (PENTAXIM™ ) and recombinant Hepatitis B (ENGERIX® PEDIATRIC) vaccines. One dose each at 2, 3, and 4 months of age.
  Interventions: Biological: DTaP-IPV//PRP~T combined; Biological: Hepatitis B vaccine

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T vaccine — 0.5 mL, Intramuscular (IM)
  Arms: Group 1: DTaP-IPV-Hep B-PRP-T
Biological: DTaP-IPV//PRP~T combined — 0.5 mL, IM
  Other Names: PENTAXIM™
  Arms: Group 2: PENTAXIM™ and ENGERIX B® PEDIATRIC
Biological: Hepatitis B vaccine — 0.5 mL, IM
  Other Names: ENGERIX B®
  Arms: Group 2: PENTAXIM™ and ENGERIX B® PEDIATRIC

SUMMARY:
To demonstrate that the immune response to hepatitis B antigen of the DTaP-IPV-Hep B-PRP~T is non-inferior to that of the association of PENTAXIM™ and ENGERIX B® one month after a three dose (2-3-4 month) primary series.

Immunogenicity

* To assess pre- and post-primary series
* To assess pre- and post-booster series.

ELIGIBILITY:
Inclusion Criteria:

* Two-month old infants of either gender on the day of inclusion
* Born at full term of pregnancy (>=37 weeks) with a birth weight >=2.5 kg
* Informed consent form signed by the parent(s) or other legal representative(s) and an institution official other than an investigator
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroid therapy
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received since birth
* Any vaccination (except BCG) in the 4 weeks preceding the first trial vaccination
* Vaccination planned in the 4 weeks following trial vaccination
* History of documented pertussis, tetanus, diphtheria, polio, Haemophilus influenzae type b or hepatitis B infection(s) (confirmed either clinically, serologically or microbiologically)
* Known personal or maternal history of HIV, Hepatitis B or Hepatitis C seropositivity
* Previous vaccination against pertussis, tetanus, diphtheria, polio or Hib, and HB infection(s)
* Coagulopathy, thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of seizures
* Febrile (axillary temperature 37.4°C [rectal equivalent temperature >=38.0°C]) or acute illness on the day of inclusion.

Ages: 50 Days to 71 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 01 June 2006 to 18 June 2007 in 1 clinical center in Turkey.
Pre-assignment Details: A total of 310 participants who met the inclusion but non of the exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-Hep B-PRP~T: Participants received 3 vaccinations with Diphtheria (D) and tetanus (T) toxoids, acellular pertussis (2-component) (aP), recombinant Hepatitis B surface antigen (HBsAg), inactivated poliomyelitis virus (IPV), and Hemophilus influenzae type b (Hib) polysaccharide conjugated to tetanus protein (DTaP-IPV-Hep B-PRP~T), with one dose each at 2, 3, and 4 months of age (Days 0, 30, and 60).
- PENTAXIM™ and ENGERIX®: Participants received 3 vaccinations with DTaP-IPV-PRP~T (PENTAXIM™ ) and recombinant Hepatitis B (ENGERIX® PEDIATRIC) vaccines, with one dose each at 2, 3, and 4 months of age (Days 0, 30, and 60).
Period: Overall Study
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX®
Started | 155 | 155
Completed | 152 | 150
Not Completed | 3 | 5
Not completed — Protocol Violation | 2 | 4
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX® | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 155 | 155 | 310
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.08 (0.090) | 2.08 (0.102) | 2.08 (0.096)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 139
  Male | 88 | 83 | 171
Region of Enrollment [Number; unit: Participants]
  Turkey | 155 | 155 | 310

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Anti HBs Seroprotection After the 3 Dose Primary Vaccination Series With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ + ENGERIX B® Vaccines
Description: Antibodies to hepatitis B surface antigen (HBs) were measured by means of automated enhanced chemoluminescence assay. Seroprotection was defined as a titer ≥ 10 mIU/mL.
Time Frame: Day 90 post first dose
Population: Seroprotection against HBs was assessed in all participants who did not have any protocol violation that might have interfered with the primary criteria evaluation (Per-Protocol Population). Totals are number of participants with available data for the endpoint.
Measure: Number; unit: Percentage of Participants
Groups:
- PENTAXIM™ and ENGERIX® PEDIATRIC: Participants received 3 vaccinations with DTaP-IPV-PRP~T (PENTAXIM™ ) and recombinant Hepatitis B (ENGERIX® PEDIATRIC) vaccines, with one dose each at 2, 3, and 4 months of age (Days 0, 30, and 60).
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX® PEDIATRIC
Number analyzed (Participants) | 134 | 128
Percentage of Participants | 94 | 96 [0 to 0]

2. Secondary Outcome: Percentage of Participants With Seroprotection Against Hepatitis B Surface Antigen, Polyribosyl Ribitol Phosphate, Diptheria, and Tetanus After the 3 Dose Primary Series With Either DTaP-IPV-Hep B-PRP~T or PENTAXIM™ + ENGERIX B®
Description: Antibodies to hepatitis B surface antigen (HBs) were measured by means of automated enhanced chemoluminescence assay. Antibodies to Polyribosyl ribitol phosphate and tetanus were measured by enzyme linked immunosorbent assay (ELISA), and antibodies to diphtheria were measured by a neutralization test using crystal violet. Seroprotection was defined as: titers ≥ 100 mIU/mL for HBs; ≥ 0.01 and ≥ 0.1 IU/mL for anti-Tetanus and anti-diphtheria, and ≥ 0.15 µg/mL and ≥ 1.0 µg/mL for anti-PRP.
Time Frame: Day 90 post first dose
Population: Seroprotection was assessed in all participants who did not have any protocol violation that might have interfered with the primary criteria evaluation (Per-Protocol Population). Totals are number of participants with available data for the endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX®
Number analyzed (Participants) | 145 | 141
Percentage of Participants
  Anti-HBs (≥ 100 mIU/mL; N = 134, 128) | 65 | 78 [0 to 0]
  Anti-PRP (≥ 0.15 µg/mL; N = 140, 138) | 91 | 98 [0 to 0]
  Anti-PRP (≥ 1.0 µg/mL; N = 140, 138) | 73 | 77 [0 to 0]
  Anti-Diphtheria (≥0.01 IU/mL; N = 144, 138) | 99 | 97 [0 to 0]
  Anti-Diphtheria (≥0.1 IU/mL; N=144, 138) | 34 | 44 [0 to 0]
  Anti-Tetanus (≥0.01 IU/mL; N = 145, 139) | 100 | 100 [0 to 0]
  Anti-Tetanus (≥0.1 IU/mL; N = 145, 139) | 100 | 99 [0 to 0]

3. Secondary Outcome: Percentage of Participants With Seroprotection Against Poliovirus Antigens After the 3 Dose Primary Series Vaccination With Either DTaP-IPV-HB-PRP~T or PENTAXIM™ + ENGERIX B®
Description: Antibodies to poliovirus types 1, 2, and 3 were measured by microneutralization on Vero cell culture. Seroprotection was defined as titers ≥8 1/dil.
Time Frame: Day 90 post first dose
Population: Anti poliovirus antibodies were assessed in all participants who did not have any protocol violation that might have interfered with the primary criteria evaluation (Per-Protocol Population). Totals are number of participants with available data for the endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX®
Number analyzed (Participants) | 145 | 141
Percentage of Participants
  Anti-Polio 1 (N = 87, 94) | 98 | 98 [0 to 0]
  Anti-Polio 2 (N = 75, 83) | 95 | 94 [0 to 0]
  Anti-Polio 3 (N = 76, 78) | 97 | 100 [0 to 0]

4. Secondary Outcome: Percentage of Participants With Anti-Pertussis Seroconversion After the 3 Dose Primary Series Vaccination With Either DTaP-IPV-HB-PRP~T or PENTAXIM™ + ENGERIX B®
Description: Antibodies to pertussis toxoid (PT) and filamentous hemagglutinin (FHA) were measured by means of enzyme linked immunosorbent assay (ELISA). Seroconversion was defined as a ≥ 4-fold increase in titer between baseline (Day 0 pre-vaccination and Day 30 post-dose 3 (Day 90).
Time Frame: Day 0 (pre-vaccination) and Day 30 post-dose 3
Population: Anti-pertussis antibodies were assessed in all participants who did not have any protocol violation that might have interfered with the primary criteria evaluation (Per-Protocol Population). Totals are number of participants with available data for the endpoint.
Measure: Number; unit: Percentage of Participants
Groups:
- DTaP-IPV-HB-PRP~T: Participants received 3 vaccinations with Diphtheria (D) and tetanus (T) toxoids, acellular pertussis (2-component) (aP), recombinant Hepatitis B surface antigen (HBsAg), inactivated poliomyelitis virus (IPV), and Hemophilus influenzae type b (Hib) polysaccharide conjugated to tetanus protein (DTaP IPV Hep B PRP T), with one dose each at 2, 3, and 4 months of age (Days 0, 30, and 60).
- PENTAXIM™ and ENGERIX®: Participants received 3 vaccinations with DTaP IPV PRP T (PENTAXIM™ ) and recombinant Hepatitis B (ENGERIX®) vaccines, with one dose each at 2, 3, and 4 months of age (Days 0, 30, and 60).
Arm/Group | DTaP-IPV-HB-PRP~T | PENTAXIM™ and ENGERIX®
Number analyzed (Participants) | 145 | 141
Percentage of Participants
  Anti-PT (Pre-dose 1; N = 143, 140) | 55 | 48 [0 to 0]
  Anti-PT (Post-dose 3; N = 143, 140) | 100 | 100 [0 to 0]
  Anti-FHA (Pre-dose 1; N = 145, 140) | 65 | 62 [0 to 0]
  Anti-FHA (Post-dose 3; N = 144, 137) | 100 | 100 [0 to 0]

5. Secondary Outcome: Geometric Mean Titers of Antibodies After the 3 Dose Primary Series With Either DTaP-IPV-HB-PRP~T or PENTAXIM™ + ENGERIX B®
Description: Antibodies to hepatitis B surface antigen (HBs) were measured by means of automated enhanced chemoluminescence assay. Antibodies to PRP, tetanus, pertussis toxoid (PT), and filamentous hemagglutinin (FHA) were measured by enzyme linked immunosorbent assay (ELISA), and antibodies to diphtheria were measured by a neutralization test using crystal violet.
Time Frame: Day 90 (30 Days post-dose 3)
Population: Geometric Mean Titers were assessed in all participants who did not have any protocol violation that might have interfered with the primary criteria evaluation (Per-Protocol Population). Totals are number of participants with available data for the endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV-HB-PRP~T | PENTAXIM™ and ENGERIX®
Number analyzed (Participants) | 145 | 141
Titers
  Anti-HBs (N = 134, 128) | 149 [115 to 191] | 265 [205 to 342]
  Anti-PRP (N = 140, 138) | 2.12 [1.62 to 2.77] | 2.37 [1.91 to 2.94]
  Anti-Diphtheria (N = 144, 138) | 0.071 [0.060 to 0.084] | 0.091 [0.075 to 0.110]
  Anti-Tetanus (N = 145, 139) | 0.839 [0.731 to 0.962] | 0.709 [0.625 to 0.804]
  Anti-Polio 1 (N = 87, 94) | 102 [74.9 to 138] | 112 [85.4 to 147]
  Anti-Polio 2 (N = 75, 83) | 73.5 [52.9 to 102] | 78.2 [58.2 to 105]
  Anti-Polio 3 (N = 76, 78) | 133 [93.0 to 190] | 214 [159 to 288]
  Anti-PT (N = 143, 140) | 123 [109 to 139] | 138 [122 to 155]
  Anti-FHA (N = 144, 137) | 102 [90.4 to 114] | 69.3 [62.0 to 77.6]

6. Secondary Outcome: Number of Participants With at Least a Solicited Injection Site or Systemic Reaction After Vaccination With Either DTaP-IPV-HB-PRP~T or PENTAXIM™ + ENGERIX B®
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, Irritability
Time Frame: Day 0 to Day 7 post any dose
Population: Solicited reactions were assessed in all participants who received at least 1 injection of study vaccine (Safety Analysis Set) according to the vaccine actually received.
Measure: Number; unit: Participants
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX®
Number analyzed (Participants) | 153 | 152
Participants
  Injection site Pain Post-dose 1 (N = 153, 152) | 70 | 55 [0 to 0]
  Injection site Pain Post-dose 2 (N = 152, 150) | 66 | 58 [0 to 0]
  Injection site Pain Post-dose 3 (N = 152, 150) | 57 | 48 [0 to 0]
  Injection site Erythema Post-dose 1 (N = 153, 152) | 23 | 17 [0 to 0]
  Injection site Erythema Post-dose 2 (N = 152, 150) | 25 | 17 [0 to 0]
  Injection site Erythema Post-dose 3 (N = 152, 150) | 30 | 17 [0 to 0]
  Injection site Swelling Post-dose 1 (N = 153, 152) | 21 | 16 [0 to 0]
  Injection site Swelling Post Dose 2 (N=152, 150) | 21 | 12 [0 to 0]
  Injection site Sweling Post Dose 3 (N = 152, 150) | 17 | 11 [0 to 0]
  Pyrexia Post-dose 1 (N = 153, 152) | 15 | 12 [0 to 0]
  Pyrexia Post-dose 2 (N = 152, 150) | 33 | 23 [0 to 0]
  Pyrexia Post-dose 3 (N = 152, 150) | 41 | 24 [0 to 0]
  Vomiting Post-dose 1 (N = 153, 152) | 57 | 44 [0 to 0]
  Vomiting Post-dose 2 (N = 152, 150) | 55 | 48 [0 to 0]
  Vomiting Post-dose 3 (N = 152, 150) | 44 | 40 [0 to 0]
  Crying Post-dose 1 (N = 153, 152) | 51 | 41 [0 to 0]
  Crying Post-dose 2 (N = 152, 150) | 54 | 38 [0 to 0]
  Crying Post-dose 3 (N = 152, 150) | 45 | 30 [0 to 0]
  Somnolence Post-dose 1 (N = 153, 152) | 51 | 45 [0 to 0]
  Somnolence Post-dose 2 (N = 152, 150) | 35 | 38 [0 to 0]
  Somnolence Post-dose 3 (N = 152, 150) | 26 | 36 [0 to 0]
  Anorexia Post-dose 1 (N = 153, 152) | 43 | 27 [0 to 0]
  Anorexia Post-dose 2 (N = 152, 150) | 48 | 35 [0 to 0]
  Anorexia Post-dose 3 (N = 152, 150) | 42 | 40 [0 to 0]
  Irritability Post-dose 1 (N = 153, 152) | 83 | 67 [0 to 0]
  Irritability Post-dose 2 (N = 152, 150) | 81 | 74 [0 to 0]
  Irritability Post-dose 3 (N = 152, 150) | 71 | 64 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed following the administration first dose of study vaccine (Day 0) through 6 months after the last dose.
Arm/Group | DTaP-IPV-Hep B-PRP~T | PENTAXIM™ and ENGERIX®
Serious Adverse Events (participants affected / at risk) | 2/153 | 3/152
Other Adverse Events (participants affected / at risk) | 83/153 | 74/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T (N=153) | PENTAXIM™ and ENGERIX® (N=152)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DTaP-IPV-Hep B-PRP~T (N=153) | PENTAXIM™ and ENGERIX® (N=152)
Vomiting (Gastrointestinal disorders) | 57 (57) | 48 (48)
Injection Site Pain (General disorders) | 70 (70) | 58 (58)
Injection Site Erythema (General disorders) | 30 (30) | 17 (17)
Injection Site Swelling (General disorders) | 21 (21) | 16 (16)
Irritability (General disorders) | 83 (83) | 74 (74)
Pyrexia (General disorders) | 41/152 (41) | 24 (24)
Anorexia (Metabolism and nutrition disorders) | 48 (48) | 40 (40)
Somnolence (Nervous system disorders) | 51 (51) | 45 (45)
Crying (Psychiatric disorders) | 54 (54) | 41 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications